CLINICAL TRIAL: NCT05342428
Title: A Phase Ⅰb, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety and Pharmacokinetics of TLL-018 in Subjects With Moderate to Severe Plaque Psoriasis
Brief Title: Safety and Efficacy of TLL018 in Patients With Plaque Psoriasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hangzhou Highlightll Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: TLL018-203
Record Dates: First submitted 2022-04-07; First posted 2022-04-22 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-07

CONDITIONS: Moderate to Severe Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): TLL018 tablets, 1piece,BID
  Interventions: Drug: TLL018 tablets
- Cohort 2 (Experimental): TLL018 tablets, 2pieces, BID
  Interventions: Drug: TLL018 tablets
- Cohort 3 (Experimental): TLL018 tablets, 3pieces, BID
  Interventions: Drug: TLL018 tablets
- Cohort 4 (Placebo Comparator): TLL018 placeboes, 3pieces, BID
  Interventions: Drug: TLL018 tablets

INTERVENTIONS:
Drug: TLL018 tablets — Oral tablets administered at different doses BID daily for 12 weeks.
  Other Names: TLL018 Placeboes

SUMMARY:
This study is a randomized, double-blind, placebo-controlled, multicenter clinical trial of about 70 subjects with moderate to severe plaque psoriasis.

DETAILED DESCRIPTION:
Successfully screened subjects will be randomized in a ratio of 2:2:2:1 and stratified to previous biologics use for psoriasis.

After a 4-week screening period (day -28-0), subjects will be randomly assigned to treatment for 12 weeks.

Clinical psoriasis area and severity index (PASI), Physician's Global Assessment (PGA), dermatological Quality of Life Index (DLQI), physical exams and Laboratory tests will be performed at baseline, the end of weeks 4, 8 and 12 respectively.

ELIGIBILITY:
Inclusion Criteria:

* Have had a diagnosis of moderate to severe plaque psoriasis for at least 6 months prior to Baseline;
* Subjects with moderate to severe plaque psoriasis covering ≥10% BSA, with a PASI ≥12 and sPGA score ≥3 at Baseline;
* Able and willing to give written informed consent.

Exclusion Criteria:

* Other types of psoriasis (such as erythrodermic psoriasis, pustular psoriasis, guttate psoriasis, etc.);
* Current drug-induced psoriasis, e.g., a new onset of psoriasis or an exacerbation of psoriasis induced by beta blockers, calcium channel blockers, antimalarial drugs or lithium;
* History or symptoms of malignancy in any organ system regardless of treatment, and regardless of evidence of recurrence or metastasis;
* Any uncontrolled clinically significant laboratory abnormality that would affect interpretation of study data or the subject's participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2022-06-10 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
treatment-emergent adverse events (AEs), serious adverse events (SAEs) and discontinuation due to AEs/SAEs | From day 1 to Weeks 12
  Number of participants with treatment-emergent adverse events (AEs), serious adverse events (SAEs) and discontinuation due to AEs/SAEs
adverse events (AEs) according to severity | From day 1 to Weeks 12
  Number of adverse events (AEs) according to severity
blood pressure from baseline | From day 1 to Weeks 12
  Change of blood pressure from baseline
pulse rate from baseline | From day 1 to Weeks 12
  Change of pulse rate from baseline
respiratory rate from baseline | From day 1 to Weeks 12
  Change of respiratory rate from baseline
temperature from baseline | From day 1 to Weeks 12
  Change of oral temperature from baseline
clinical laboratory abnormalities compared to baseline | From day 1 to Weeks 12
  Number of participants with clinical laboratory abnormalities compared to baseline
ECG parameters from baseline | From day 1 to Weeks 12
  Change in 12-lead electrocardiogram (ECG) parameters (PR Interval, QRS Complex, QT Interval, QTC Interval) from baseline
physical examination findings from baseline | From day 1 to Weeks 12
  Number of participants with changes in physical examination findings from baseline
Cmax of TLL018 | 0 hour (pre-dose - within 30 minutes prior to dosing), and at 0.5, 1, 2, 4 and 12 hours post-dose
  Maximum observed plasma concentration (Cmax) of TLL018

SECONDARY OUTCOMES:
PASI score decreased from baseline at week 4 | Baseline to Week 4
  The percentage of subjects whose PASI score decreased by at least 50%(PASI 50) 75%(PASI 75) 90%(PASI 90) and 100%(PASI 100) from baseline at week 4 when comparing TLL-018 with placebo
PASI score decreased from baseline at week 8 | Baseline to Week 8
  The percentage of subjects whose PASI score decreased by at least 50%(PASI 50) 75%(PASI 75) 90%(PASI 90) and 100%(PASI 100) from baseline at week 8 when comparing TLL-018 with placebo
PASI score decreased from baseline at week 12 | Baseline to Week 12
  The percentage of subjects whose PASI score decreased by at least 50%(PASI 50) 75%(PASI 75) 90%(PASI 90) and 100%(PASI 100) from baseline at week 12 when comparing TLL-018 with placebo
(sPGA) 0/1 response at week 4 | Baseline to Weeks 4
  static Physician Global Assessment (sPGA) 0/1 response
(sPGA) 0/1 response at week 8 | Baseline to Weeks 8
  static Physician Global Assessment (sPGA) 0/1 response
(sPGA) 0/1 response at week 12 | Baseline to Weeks 12
  static Physician Global Assessment (sPGA) 0/1 response

CONTACTS AND LOCATIONS:
Locations (1):
- 88 Jiefang Road, Shangcheng District, Hangzhou City, Zhejiang Province, Hangzhou, Zhejiang, China